CLINICAL TRIAL: NCT00202800
Title: Phase II Trial to Evaluate Gemcitabine and Etoposide for Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Van Andel Research Institute (Other); Eli Lilly and Company (Industry); Battle Creek Health System (Other); Mercy Health System (Network); Metropolitan Hospital, Michigan (Other); Mecosta County General Hospital (Unknown); Munson Medical Center (Other); Saint Mary's Health Network (Other)
Responsible Party: Marianne Lange, MD, Spectrum Health
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VARI-002-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Gemcitabine/Etoposide; Ras-mutation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Etoposide

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: Gemcitabine, Etoposide — Pancreatic cancer is a devastating disease. Previous research shows a correlation between a specific oncogene change (ras-mutation) and enhanced sensitivity to two chemotherapy drugs combined: gemcitabine and etoposide. This Phase II trial will evaluate this drug combination for locally advanced and metastatic pancreatic cancer

SUMMARY:
Pancreatic cancer is a devastating disease. Previous research shows a correlation between a specific oncogene change (ras-mutation) and enhanced sensitivity to two chemotherapy drugs combined: gemcitabine and etoposide. This Phase II trial will evaluate this drug combination for locally advanced and metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This is a Phase II single-armed study evaluating potential benefits of the gemcitabine and etoposide combination in the treatment of patients with locally advanced or metastatic pancreatic cancer. The study will involve approximately 30-40 adult patients with pancreatic cancer. Response rate, duration of response, overall survival, quality of life and toxicity associated with the combination therapy will be evaluated.

Primary Objective To evaluate the response rate of patients with histologically or cytologically confirmed pancreatic cancer, previously untreated with chemotherapy with the exception of 5FU given as part of an adjuvant regimen, who receive the gemcitabine-etoposide combination therapy.

Secondary Objectives 1. To evaluate the duration of response in the defined study population. 2. To evaluate the overall survival. 3. To evaluate the quality of life associated with this treatment combination.4.To describe the toxicity profile. 5.To collect clinical specimens from the defined study population for the evaluation of potential molecular correlates of diagnosis, disease progression, treatment outcomes, survival, and/or treatment-associated toxicity by proteomics and microarray technologies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic adenocarcinoma of the pancreas.
* Patients may have received prior immunotherapy, radiation therapy, or surgery, but must be > 4 weeks out from therapy and have recovered fully from its effects.
* Patients must be 18 years of age or older.
* Patients must have unidimensional measurements obtainable using RECIST criteria (see Protocol Attachment E).
* Karnofsky Performance Scale must be 50 or better (see Protocol Attachment A).
* Patient must have the following hematologic and chemical parameters:

  * ANC > 1,000 cells/mm3
  * Hemoglobin > 9 gm/dL
  * Platelets > 100,000 cells/mm3
  * SGOT/SGPT < 3 x normal, unless there is known liver involvement. Then they must be < 5x normal.
  * Bilirubin < 2.0 mg/dL
  * Creatinine < 2.0 mg/dL
* Female within childbearing years must use an accepted contraceptive method.
* Patient must have a life expectancy of at least eight (8) weeks.
* A signed informed consent must be obtained prior to study entry.

Exclusion Criteria:

* Previous chemotherapy with the exception of 5FU given as part of an adjuvant regimen.
* Pregnant or nursing females.
* Concurrent radiation therapy.
* Patients with other active neoplasms are ineligible.
* Patients with serious active infections or other underlying medical conditions, which would impair their ability to receive the treatment as prescribed.

Disease Diagnostic Criteria and Staging:

* Patients must have a histologic or cytologic diagnosis of locally advanced or metastatic adenocarcinoma of the pancreas using standard pathologic criteria.
* Staging will be according to AJCC criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2002-03; Primary Completion 2007-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate | study completion

SECONDARY OUTCOMES:
To evaluate the duration of response | study completion
To evaluate the overall survival | study completion
To evaluate the quality of life | study completion
To describe the toxicity profile | study completion

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Lange, MD, Principal Investigator — Grand Rapids Clinical Oncology Program
Locations (1):
- Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan, United States